CLINICAL TRIAL: NCT04316468
Title: Evaluation of Cardiac Strain Using Speckle Tracking Echocardiography During Orthotopic Liver Transplantation
Brief Title: Cardiac Strain Using Speckle Tracking Echocardiography During Orthotopic Liver Transplantation
Status: Terminated | Type: Observational
Why Stopped: Unable to find software to open saved images for analysis
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen Aniskevich, III, Principal Investigator, Mayo Clinic
Other Study IDs: 20-001209
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Liver Transplant Disorder; Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers are trying to improve the understanding of systolic function of the heart at the time of liver reperfusion in patients undergoing orthotopic liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Undergoing primary orthotopic liver transplantation

Exclusion Criteria:

* Redo orthotopic transplantation
* Acute or fulminant liver failure
* Patient with pre-existing atrial fibrillation or hypertrophic cardiomyopathy
* Patients with an abnormal preoperative stress test (EF <55%, areas of prior infarct, ongoing ischemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sequential liver transplant candidates (adults) will be approached for consent to participate in the study at the time of liver transplantation by a member of the liver anesthesia team.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Degree of change in cardiac strain | Up to 1 hour after graft reperfusion
  Evaluate the degree of change to cardiac strain using speckle tracking echocardiography

SECONDARY OUTCOMES:
Pattern of right and left ventricular strain | Up to 5 hours from the time of surgery start
  Describe the pattern of right and left ventricular strain throughout the course of orthotopic liver transplantion.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Aniskevich, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials